CLINICAL TRIAL: NCT05429047
Title: Priming of the NEonatal Immune System by Transfer of Maternal Immunity
Acronym: NEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NEST
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Maternal Vaccine Exposure; Respiratory Infections in Children
Keywords: first year of life; development of the immune system; antibody transfer via placenta; breast milk
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, PBMCs, stool, nasal secretions, breast milk, nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SARS-CoV-2 vaccine during pregnancy: Pregnant women who received a vaccine against SARS-CoV-2 during pregnancy and their children
  Interventions: Biological: Tozinameran
- SARS-CoV-2 infection during pregnancy: Pregnant women who were diagnosed with a SARS-CoV-2 infection during pregnancy and their children
  Interventions: Other: COVID-19
- SARS-CoV-2 vaccine or infection before pregnancy: Pregnant women who neither received a COVID-19 vaccine nor were diagnosed with COVID-19 during their pregnancy but had either a COVID-19 vaccine or infection before pregnancy and their children
  Interventions: Other: No SARS-CoV-2 exposure
- No exposure: Pregnant women, who were never exposed to a SARS-CoV-2 vaccine or infection until the birth and their children
  Interventions: Other: No SARS-CoV-2 exposure

INTERVENTIONS:
Biological: Tozinameran — Tozinameran during pregnancy
  Groups: SARS-CoV-2 vaccine during pregnancy
Other: COVID-19 — SARS-CoV-2 infection during pregnancy
  Groups: SARS-CoV-2 infection during pregnancy
Other: No SARS-CoV-2 exposure — No SARS-CoV-2 exposure during pregnancy
  Groups: No exposure; SARS-CoV-2 vaccine or infection before pregnancy

SUMMARY:
Newborn babies and infants are susceptible to infections as their immune system is still immature. Maternal immune factors for example antibodies and immune cells mitigate this vulnerability. They are transferred from mother to child via the placenta during pregnancy or by breast milk after birth and provide protection against infectious diseases.

In the case of SARS-CoV-2 it has already been shown that specific antibodies are transferred from mother to children after infection or vaccination during pregnancy. However, to this date it is not known how long such an antibody-mediated protection lasts in children and if this "passive" immunity actually protects infants from SARS-CoV-2 infection in the first months of life.

In general, there is still little knowledge about the influence of maternal infections during pregnancy, transfer of maternal immune factors to the child and development of the child's immune system and health in the first months of life.

Here, the investigators aim to study transferred immunity (i.e. specific antibodies) against SARS-CoV-2 in children of mothers who received a SARS-CoV-2 vaccination during pregnancy or had a SARS-CoV-2 infection during pregnancy with mothers not exposed or exposed before pregnancy.

In addition, the investigators will comprehensively characterize the development of the cellular immune system in the first year of life (umbilical cord blood, age 6 and 12 months) to explore how maternal exposure to infectious diseases or vaccines influences the development of the immune system of the newborn infant.

DETAILED DESCRIPTION:
Pregnant women are at increased risk of severe SARS-CoV-2 infections including ARDS and multi-organ failure and increased risk of miscarriages or premature birth. Although pregnant women were not included in market authorization studies, inoculation with mRNA based vaccines is now recommended in Germany.

Vertical transmission rate of SARS-CoV-2 of infected mothers is < 5% and newborns present in the majority of cases with mild symptoms only. Overall, morbidity and mortality of SARS-CoV-2 infections in childhood are significantly lower in children than adults however it is higher in young infants in the first year of life. Further research into the disease burden of SARS-CoV-2 in neonates and young infants and preventative strategies regarding maternal vaccination strategies is therefore urgently needed.

Pregnant women show robust antibody responses to both mRNA vaccines as well as infection including IgG against spike protein, neutralizing antibodies and spike-specific T cell responses. Both spike-protein IgG as well as neutralizing antibodies can be found in cord blood after vaccination and antibody levels can be detected in the child for up to at least 2-3 months. Equally, vaccination of lactating mothers results in transfer of spike-protein reactive secretory IgA and T cells.

Although there is generally good proof of passive transfer of antibodies to the unborn child and neonate transplacentally and via mother's milk, many open question remain. It remains unclear, which vaccination regime results in optimal transfer to the newborn child, if vaccination shows improved protection to infection or if general boostering should be recommended for all women in the second trimenon irrespective of previous vaccination or infection history. Additionally, most studies showing vertical transfer of antibodies to the newborn child have been done with small numbers of mother-child dyads and without clinical follow-up regarding risk of SARS-CoV-2 infection in the first year of life.

Furthermore, it remains unexplored if maternal SARS-CoV2 infection or vaccination during pregnancy shapes the fetus immune system with long-lasting effects. Maternal infections can shape the neonatal immune system even if the fetus remains uninfected. Similar effects have been suggested for maternal vaccination during pregnancy. Studies investigating the effect of maternal SARS-CoV-2 infection during pregnancy on uninfected neonates show mild cytokine response in the neonate as measured in cord blood but no major alterations to lymphocyte subsets and T cell repertoire. However, comprehensive immunophenotyping of the newborns' cellular immune system after either SARS-CoV-2 infection and/ or vaccination during pregnancy with clinical follow-up of the children in the first year of life has not been done yet.

With this study, the investigators aim to examine the antibody response in mother-child dyads after either SARS-CoV-2 vaccination or infection during pregnancy compared to mothers with SARS-CoV-2 vaccination or infection before pregnancy. Antibody titers will be measured in the blood of children and mothers as well as mother's milk.

This data will be combined with comprehensive phenotyping of the cellular immune cells, microbiome analysis and data regarding the child's clinical outcome regarding respiratory infections in the first year of life.

ELIGIBILITY:
Inclusion Criteria:

For mothers:

* ≥ 18 years
* Informed Consent

For children:

- Informed Consent of the parents

Exclusion Criteria:

During pregnancy:

* Premature rupture of membranes (>48h before delivery)
* Preterm Birth (<32+0 weeks of pregnancy)
* Preeclampsia, HELLP syndrome and Eclampsia
* Twin-to-twin transfusion syndrome
* Hydrops fetalis
* Oncological disease of the mother
* Immunodeficiency, autoimmune or immunological disorder of the mother
* Further health conditions of mother or fetus that may influence the results of the study according to the opinion of the study team

In children after delivery:

* Delivery >48h after rupture of membranes
* Perinatal asphyxia (APGAR score at 10 minutes: < 5 and/or blood acidosis (fetal umbilical artery pH: < 7.0, arterial base deficit ≥ 12 mmol/L))
* High flow therapy or non-invasive or invasive ventilation after birth
* Treatment with vasopressors or inotropes after birth
* Treatment with intravenous antibiotics after birth
* Neonatal jaundice with need for an exchange transfusion
* Postnatal need for blood transfusions
* Further health conditions of the child that may influence the results of the study according to the opinion of the study team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women recruited from the Department of Obstetrics and Gynecology, Hannover Medical School
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
anti-SARS-CoV-2 IgG Titer and neutralizing antibody titers in cord blood | at delivery

SECONDARY OUTCOMES:
anti-SARS-CoV-2 IgG titer and neutralizing antibody titers in maternal blood | at delivery, 6 months after delivery, 12 months after delivery
anti-SARS-CoV-2 IgG titer and neutralizing antibody titers in peripheral blood of the child | at 6 months of life, at 12 months of life
anti-SARS-CoV-2 IgG/IgA titer and neutralizing antibody titers in breast milk | first week after delivery, 6 month after delivery
SARS-CoV-2 specific T cells in cord blood | at delivery
SARS-CoV-2 specific T cells immunity in maternal blood | at delivery
SARS-CoV-2 specific T cells in peripheral blood of the child | at 6 months of life, at 12 months of life
SARS-CoV-2 specific T cells in breast milk | first week after delivery, 6 month after delivery
total IgG in cord blood and maternal blood | at delivery
COVID-19 infection rate in children | first year of life

OTHER OUTCOMES:
Comprehensive Immunophenotyping of blood leukocytes | At delivery (cord blood), 6 months, 12 months
  spectral flow cytometry
Rates of bacterial phyla in samples from gastrointestinal and respiratory tract | 3rd day of life, 6 months, 12 months
  Microbiome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gesine Hansen, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School (Medizinische Hochschule Hannover, MHH), Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No